CLINICAL TRIAL: NCT00957658
Title: Accolade® TMZF® Study A Prospective, Post-market, Non-randomized, Multi-center Evaluation of the Accolade® TMZF® Hip Stem
Brief Title: Accolade® TMZF® Hip Stem Outcomes Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stryker Orthopaedics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 59
Record Dates: First submitted 2009-08-10; First posted 2009-08-12 (Estimated); Results first posted 2014-08-15 (Estimated); Last update posted 2017-08-14 (Actual); Status verified 2016-07

CONDITIONS: Arthroplasty, Replacement, Hip
Keywords: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Accolade® TMZF® Hip Stem (Other): Accolade® TMZF® Hip Stem Study Device
  Interventions: Device: Accolade® TMZF® Hip Stem

INTERVENTIONS:
Device: Accolade® TMZF® Hip Stem — Accolade® TMZF® Hip Stem

SUMMARY:
The purpose of this study is to evaluate clinical and radiographic outcome data in patients implanted with the Accolade® TMZF® femoral stem.

DETAILED DESCRIPTION:
A prospective, post-market, multi-centered clinical evaluation of the Accolade® TMZF® hip stem device. All patients enrolled will receive the study device. All study patients will undergo a preoperative central Dual energy X-ray absorptiometry (DXA) scan to determine bone mineral density (BMD) values.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is a candidate for a primary total hip replacement.
2. Patient has primary diagnosis of osteoarthritis (OA).
3. Male and non-pregnant female patients ages 18 to 90.
4. Patient has signed an Institutional Review Board (IRB) approved, study specific Informed Patient Consent Form.
5. Patient willing and able to comply with postoperative scheduled clinical and radiographic evaluations and rehabilitation.
6. Patient capable of undergoing a pre-op central DXA (dual-energy x-ray absorptiometry) scan for a bone mineral density (BMD) reading.

Exclusion Criteria:

1. Patient has an active infection within the affected hip joint.
2. Patient requires a revision surgery of a previously implanted total hip arthroplasty or hip fusion to the affected joint.
3. Patient who is morbidly obese, Body Mass Index (BMI) > 40.
4. Patient has a neuromuscular or neurosensory deficiency, which limits ability to evaluate the safety and efficacy of the device.
5. Patient has the following diagnosed systemic diseases: Paget's disease, renal osteodystrophy, lupus erythematosus, rheumatoid arthritis, metabolic bone disease and sickle cell anemia.
6. Patient is immunologically suppressed or receiving chronic steroids more than 30 days. Patients receiving oral or IV steroids within one month of surgery.
7. Patient is a prisoner.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2006-03; Primary Completion 2011-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Krushell, MD, Study Chair — Baystate Medical Center; Carlton Savory, MD, Principal Investigator — Hughston Sports Medicine Center; Robert Zann, MD, Principal Investigator — Boca Raton Community Hospital; Steven Gausewitz, MD, Principal Investigator — Hoag Hospital; R. Scott Oliver, MD, Principal Investigator — Jordan Hospital; Mary O'Connor, MD, Principal Investigator — Mayo Clinic; Anthony Sanchez, MD, Principal Investigator — Spartanburg Regional Health Service District, Inc; Mark Visk, MD, Principal Investigator — Spartanburg Regional Health Service District, Inc; Steven Teeny, MD, Principal Investigator — St. Clare Hospital; Alan Valadie, MD, Principal Investigator — Coastal Orthopedics and Sports Medicine; Steven Zelicof, MD, Principal Investigator — Sound Shore Medical Center of Westchester; James Bates, MD, Principal Investigator — Alvarado Hospital
Locations (11):
- United States (11):
  - Newport Orthopaedic Institute, Newport Beach, California
  - Alvarado Ortho Medical Group, San Diego, California
  - Orthopaedic Surgery Associates, Boynton Beach, Florida
  - Coastal Orthopaedics, Bradenton, Florida
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Hughston Clinic P.A., Columbus, Georgia
  - Plymouth Bay Ortho Association, Duxbury, Massachusetts
  - New England Orthopaedic Surgeons, Springfield, Massachusetts
  - Specialty Orthopaedics, Harrison, New York
  - Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Northwest Orthopaedic Institute, Tacoma, Washington

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 241 participants/249 hips - 7 censored participants/7 hips = 234 participants/242 hips
Groups:
- Accolade® TMZF® Hip Stem: Accolade® TMZF® Hip Stem Study Device. Participants have one or both hips replaced. If both hips were replaced, but only one hip completed the primary endpoint, the participant is counted as completed.
Period: Overall Study
Arm/Group | Accolade® TMZF® Hip Stem
Started | 234
Completed | 169 (Completed/Not completed counts are based on participant status at the 2yr primary outcome interval.)
Not Completed | 65
Not completed — Death | 1
Not completed — Lost to Follow-up | 4
Not completed — Withdrawal by Subject | 12
Not completed — Revision | 1
Not completed — Incomplete 2 yr data | 28
Not completed — Site termination | 10
Not completed — unwilling/unable to return | 2
Not completed — surgery cancelled | 2
Not completed — Protocol Violation | 5

BASELINE CHARACTERISTICS:
Population: Participants who were censored protocol violations or who were enrolled but did not have surgery or age data was not available, are not included in the baseline analysis.
Arm/Group | Accolade® TMZF® Hip Stem
Number analyzed (Participants) | 234
Age, Continuous [Mean (Standard Deviation); unit: years] — 1. Age results are based on 226 participants as there were 8 participants missing age data.
  2. For bilateral total hip replacement participants, the age at the time of the initial hip surgery is used.
  years | 68.94 (9.77)
Sex/Gender, Customized [Number; unit: participants] — Gender is based on 229 participants as there were 5 participants missing gender data.
  participants
    Female | 149
    Male | 80
Region of Enrollment [Number; unit: participants]
  United States | 234

OUTCOME MEASURES:

1. Primary Outcome: Combined Percentage (%) Cases Without Aseptic Loosening, Intraoperative Femoral Fracture or Thigh Pain
Time Frame: 2 years
Measure: Number; unit: percentage of hips
Units Other Than Participants: hips
Arm/Group | Accolade® TMZF® Hip Stem
Number analyzed (Participants) | 169
Number analyzed (hips) | 174
percentage of hips | 98.85
Statistical Analysis 1: Comparison: Accolade® TMZF® Hip Stem; Literature control = 96% with no aseptic loosening, intraop femoral fracture or thigh pain at 2 years; Test type: Non-Inferiority or Equivalence — Non-inferiority margin = 6%; p < .0001, Asymptotic WALD test

2. Secondary Outcome: Percentage (%) of Hip Stems With Aseptic Loosening
Description: Aseptic loosening is defined as a continuous radiolucency that surrounds the entire femoral stem porous coating-bone interface and that measures greater than 2 mm in thickness, and 5 mm or more of stem subsidence. Continuous radiolucency must be present in Zones 1, 2, 6 and 7 of the AP radiographic view and/or present in Zones 8, 9, 13 and 14 of the M/L radiographic view.
Time Frame: 5 years
Population: Participants with available data: 111 hips in 106 participants had a radiographic evaluation at 5 years.
Measure: Number; unit: percentage of hips
Units Other Than Participants: hips
Groups:
- Accolade® TMZF® Hip Stem: Subjects who received the Accolade® TMZF® Hip Stem
Arm/Group | Accolade® TMZF® Hip Stem
Number analyzed (Participants) | 106
Number analyzed (hips) | 111
percentage of hips | 0

3. Secondary Outcome: Revision/Removal Rates
Description: The percentage (%) of hips with revision or removal of any total hip replacement component (acetabular cup, femoral stem or femoral head) is reported at the 2 and 5 year postoperative intervals.
Time Frame: 2 and 5 years
Population: Participants with available data: The revision/removal rate of any total hip replacement component at 2 years is reported for 182 hips/176 participants. The revision/removal rate of any component at 5 years is reported for 141 hips/136 participants.
Measure: Number; unit: percentage of hips/any component revised
Units Other Than Participants: hip
Arm/Group | Accolade® TMZF® Hip Stem
Number analyzed (Participants) | 176
Number analyzed (hip) | 182
percentage of hips/any component revised
  Revision/removal rate % at 2 years | 1.65
  Revision/removal rate % at 5 years | 2.84

4. Secondary Outcome: Change in Harris Hip Score (HHS)
Description: The change in HHS is reported by comparing the mean preoperative, 2 and 5 year postoperative scores. Scores can range from 0 to 100 with 0 being the worst and 100 being the best score. A score of 80-100 is considered good-excellent and a score of less than or equal to 79 is considered fair-poor. 90-100 = excellent, 80-89 = good, 70-79 = fair, 0-69 = poor.
Time Frame: Preoperative, 2 and 5 years
Population: Participants with available data: A total of 195 hips had a preoperative score, 174 had a 2 year score, and 117 had a 5 year score.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: hips
Arm/Group | Accolade® TMZF® Hip Stem
Number analyzed (Participants) | 189
Number analyzed (hips) | 195
units on a scale
  Mean HHS score Preoperative (n=195) | 50.1 (11.99)
  Mean HHS score 2 years (n=174) | 89.4 (12.67)
  Mean HHS score 5 years (N=117) | 92.2 (12.61)
Statistical Analysis 1: Comparison: Accolade® TMZF® Hip Stem; Improvement from preop to 2 year and preop to 5 year; Test type: Superiority or Other; p < .0001, Sign test

5. Secondary Outcome: Change in SF-12 Score
Description: The change in SF-12 is reported by comparing the mean preoperative, 2 and 5 year postoperative scores.The SF-12 Health Survey is a 12-item patient completed questionnaire to measure general health and well-being. It includes a physical and mental status component score; each ranging from 0-100. Low values represent a poor health state and high values represent a good health state.
Time Frame: Preoperative, 2 and 5 years
Population: Participants with available data: A total of 217 hips had preoperative scores, 175 had 2 year and 121 had 5 year scores.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: hips
Arm/Group | Accolade® TMZF® Hip Stem
Number analyzed (Participants) | 210
Number analyzed (hips) | 217
units on a scale
  Mean SF12 Physical Preoperative (N=217) | 32.3 (8.3)
  mean SF12 Mental Preoperative (N=217) | 49.1 (11.99)
  Mean SF12 Physical 2 years (N=175) | 45.6 (11.17)
  Mean SF12 Mental 2 years (N=175) | 54.2 (8.41)
  Mean SF-12 Physical 5 years (N=121) | 44.8 (10.62)
  Mean SF-12 Mental 5 years (N=121) | 53.4 (9.45)
Statistical Analysis 1: Comparison: Accolade® TMZF® Hip Stem; Compare Pre-op SF-12 Physical Score preop to 2 year and preop to 5 year; Test type: Superiority or Other; p < .0001, t-test, 2 sided
Statistical Analysis 2: Comparison: Accolade® TMZF® Hip Stem; Change in SF-12 Mental Score preop to 2 years; Test type: Superiority or Other; p < .0001, Sign test
Statistical Analysis 3: Comparison: Accolade® TMZF® Hip Stem; Compare SF-12 Mental Score preop to 5 years; Test type: Superiority or Other; p = .0004, t-test, 2 sided

6. Secondary Outcome: Change in Lower Extremity Activity Scale (LEAS) Score
Description: The change in LEAS is reported by comparing the mean preoperative, 2 and 5 year postoperative scores.The LEAS is completed by the participant to assess activity level. Activity levels were ordered in terms of intensity from 1 to 18, with 18 indicating the highest activity level. The mean preoperative, 2 and 5 year scores are reported to assess improvement.
Time Frame: Preoperative, 2 and 5 years
Population: Participants with available data: A total of 231 hips had a preoperative score, 181 had a 2 year, and 129 had a 5 year score.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: hips
Arm/Group | Accolade® TMZF® Hip Stem
Number analyzed (Participants) | 233
Number analyzed (hips) | 231
units on a scale
  Mean LEAS Preoperative (n=231) | 8.4 (3.32)
  Mean LEAS 2 year (N=181) | 10.4 (3.18)
  Mean LEAS 5 year (N=129) | 10.2 (3.34)
Statistical Analysis 1: Comparison: Accolade® TMZF® Hip Stem; Compare LEAS score preop to 2 years and preop to 5 years; Test type: Superiority or Other; p < .0001, Sign test

7. Secondary Outcome: PEQ (Patient Expectation Questionnaire) Overall Satisfaction
Description: The PEQ is a study sponsor generated outcomes form. It is a one page questionnaire completed by the participant to assess lifestyle recovery post-surgery. Preoperatively, participants are asked to identify 3 of 12 different expectations that they most want to achieve after hip surgery. At 6 months,1 year and 2 years post-surgery participants evaluated the 3 expectations they identified and assessed their overall satisfaction and percent achievement.
  EXPECTATIONS KEY:
  Participate in recreational activities (dancing,traveling,gardening)
  Exercise or participate in sports
  Independently perform household chores/daily routine
  Easily change position,sit to stand/stand to sit
  Remove need for cane crutch or walker
  Use stairs normally step by step
  Ability to sleep through night
  Maintain social activites,caring for someone,playing with children
  Use public transportation or drive
  Maintain psychological well-being
  Maintain sexual activity
  Maintain employment
Time Frame: 6 months, 1 year and 2 years
Population: Participants with available data: A total of 206 hips had 6 month data; a total of 203 hips had 1 year data; a total of 178 hips had 2 year data. Percentage of participants who were satisfied with the result is reported for each expectation at these intervals.
Measure: Number; unit: percentage of particpants
Units Other Than Participants: hips
Arm/Group | Accolade® TMZF® Hip Stem
Number analyzed (Participants) | 201
Number analyzed (hips) | 206
percentage of particpants
  Recreation 6 mo (n=97) | 84.5
  Recreation 1 yr (n=95) | 88.4
  Recreation 2 yr (n=76) | 85.5
  Exercise/sports 6 mo (n=79) | 89.9
  Exercise/sports 1 yr (n=79) | 89.9
  Exercise/sports 2 yr (n=67) | 91
  Chores 6 mo (n=71) | 91.5
  Chores 1 yr (n=65) | 86.2
  Chores 2 yr (n=58) | 96.6
  Change position 6 mo (n=57) | 87.7
  Change position 1 yr (n=58) | 87.9
  Change position 2 yr (n=43) | 90.7
  No cane/crutch/walker 6 mo (n=57) | 94.7
  No cane/crutch/walker 1 yr (n=53) | 94.3
  No cane/crutch/walker 2 yr (n=49) | 93.9
  Stairs normally 6 mo (n=52) | 80.8
  Stairs normally 1 yr (n=58) | 86.2
  Stairs normally 2 yr (n=45) | 91.1
  Sleep 6 mo (n=52) | 71.2
  Sleep 1 yr (n=49) | 77.6
  Sleep 2 yr (n=51) | 84.3
  Maintain activities 6 mo (n=44) | 90.9
  Maintain activities 1 yr (n=41) | 87.8
  Maintain activities 2 yr (n=38) | 94.7
  Transportation 6 mo (n=27) | 96.3
  Transportation 1 yr (n=29) | 96.6
  Transportation 2 yr (n=24) | 95.8
  Well-being 6 mo (n=21) | 85.7
  Well-being 1 yr (n=20) | 95
  Well-being 2 yr (n=15) | 86.7
  Sexual activity 6 mo (n=15) | 80
  Sexual activity 1 yr (n=13) | 84.6
  Sexual activity 2 yr (n=12) | 66.7
  Employment 6 mo (n=12) | 83.3
  Employment 1 yr (n=11) | 81.8
  Employment 2 yr (n=8) | 87.5

8. Secondary Outcome: PEQ (Patient Evaluation Questionnaire) Percent Achievement
Description: as for outcome 7
Time Frame: 6 months, 1 year, 2 years
Population: Participants with available data: A total of 206 hips had 6 month data; a total of 203 hips had 1 year data; a total of 178 hips had 2 year data. Participants select 3 expectations and assess percent achievement (100%,75%,50%,25%,or 0%) at 6 mos, 1 yr and 2 yrs.
Measure: Number; unit: percentage of participants
Units Other Than Participants: hips
Arm/Group | Accolade® TMZF® Hip Stem
Number analyzed (Participants) | 201
Number analyzed (hips) | 206
percentage of participants
  Recreation 100% 6 mo (n=101) | 42.6
  Recreation 100% 1 yr (n=97) | 55.7
  Recreation 100% 2 yr (n=83) | 47.0
  Recreation 75% 6 mo (n=101) | 33.7
  Recreation 75% 1 yr (n=97) | 28.9
  Recreation 75% 2 yr (n=83) | 28.9
  Recreation 50% 6 mo (n=101) | 9.9
  Recreation 50% 1 yr (n=97) | 8.2
  Recreation 50% 2 yr (n=83) | 12.0
  Recreation 25% 6 mo (n=101) | 11.9
  Recreation 25% 1 yr (n=97) | 3.1
  Recreation 25% 2 yr (n=83) | 8.4
  Recreation 0% 6 mo (n=101) | 2.0
  Recreation 0% 1 yr (n=97) | 4.1
  Recreation 0% 2 yr (n=83) | 3.6
  Exercise/sports 100% 6 mo (n=81) | 43.2
  Exercise/sports 100% 1 yr (n=82) | 51.2
  Exercise/sports 100% 2 yr (n=74) | 44.6
  Exercise/sports 75% 6 mo (n=81) | 37.0
  Exercise/sports 75% 1 yr (n=82) | 29.3
  Exercise/sports 75% 2 yr (n=74) | 32.4
  Exercise/sports 50% 6 mo (n=81) | 9.9
  Exercise/sports 50% 1 yr (n=82) | 9.8
  Exercise/sports 50% 2 yr (n=74) | 5.4
  Exercise/sports 25% 6 mo (n=81) | 4.9
  Exercise/sports 25% 1 yr (n=82) | 8.5
  Exercise/sports 25% 2 yr (n=74) | 13.5
  Exercise/sports 0% 6 mo (n=81) | 4.9
  Exercise/sports 0% 1 yr (n=82) | 1.2
  Exercise/sports 0% 2 yr (n=74) | 4.1
  Chores 100% 6 mo (n=74) | 71.6
  Chores 100% 1 yr (n=72) | 65.3
  Chores 100% 2 yr (n=65) | 58.5
  Chores 75% 6 mos (n=74) | 14.9
  Chores 75% 1 yr (n=72) | 19.4
  Chores 75% 2 yr (n=65) | 27.7
  Chores 50% 6 mo (n=74) | 6.8
  Chores 50% 1 yr (n=72) | 5.6
  Chores 50% 2 yr (n=65) | 7.7
  Chores 25% 6 mo (n=74) | 6.8
  Chores 25% 1 yr (n=72) | 6.9
  Chores 25% 2 yr (n=65) | 6.2
  Chores 0% 6 mo (n=74) | 0
  Chores 0% 1 yr (n=72) | 2.8
  Chores 0% 2 yr (n=65) | 0
  Change position 100% 6 mo (n=63) | 58.7
  Change position 100% 1 yr (n=61) | 60.7
  Change position 100% 2 yr (n=49) | 57.1
  Change position 75% 6 mo (n=63) | 28.6
  Change position 75% 1 yr (n=61) | 31.1
  Change position 75% 2 yr (n=49) | 26.5
  Change position 50% 6 mo (n=63) | 6.3
  Change position 50% 1 yr (n=61) | 8.2
  Change position 50% 2 yr (n=49) | 14.3
  Change position 25% 6 mo (n=63) | 6.3
  Change position 25% 1 yr (n=61) | 0
  Change position 25% 2 yr (n=49) | 2.0
  Change position 0% 6 mo (n=63) | 0
  Change position 0% 1 yr (n=61) | 0
  Change position 0% 2 yr (n=49) | 0
  No cane/crutch/walker 100% 6 mo (n=58) | 79.3
  No cane/crutch/walker 100% 1 yr (n=54) | 79.6
  No cane/crutch/walker 100% 2 yr (n=53) | 77.4
  No cane/crutch/walker 75% 6 mo (n=58) | 12.1
  No cane/crutch/walker 75% 1 yr (n=54) | 7.4
  No cane/crutch/walker 75% 2 yr (n=53) | 7.5
  No cane/crutch/walker 50% 6 mo (n=58) | 1.7
  No cane/crutch/walker 50% 1 yr (n=54) | 7.4
  No cane/crutch/walker 50% 2 yr (n=53) | 7.5
  No cane/crutch/walker 25% 6 mo (n=58) | 5.2
  No cane/crutch/walker 25% 1 yr (n=54) | 5.6
  No cane/crutch/walker 25% 1 yr (n=53) | 5.7
  No cane/crutch/walker 0% 6 mo (n=58) | 1.7
  No cane/crutch/walker 0% 1 yr (n=54) | 0
  No cane/crutch/walker 0% 2 yr (n=53) | 1.9
  Stairs normally 100% 6 mo (n=56) | 51.8
  Stairs normally 100% 1 yr (n=59) | 62.7
  Stairs normally 100% 2 yr (n=47) | 55.3
  Stairs normally 75% 6 mo (n=56) | 25
  Stairs normally 75% 1 yr (n=59) | 6.8
  Stairs normally 75% 2 yr (n=47) | 8.5
  Stairs normally 50% 6 mo (n=56) | 7.1
  Stairs normally 50% 1 yr (n=59) | 18.6
  Stairs normally 50% 2 yr (n=47) | 19.1
  Stairs normally 25% 6 mo (n=56) | 8.9
  Stairs normally 25% 1 yr (n=59) | 8.5
  Stairs normally 25% 2 yr (n=47) | 10.6
  Stairs normally 0% 6 mo (n=56) | 7.1
  Stairs normally 0% 1 yr (n=59) | 3.4
  Stairs normally 0% 2 yr (n=47) | 6.4
  Sleep 100% 6 mo (n=55) | 43.6
  Sleep 100% 1 yr (n=53) | 39.6
  Sleep 100% 2 yr (n=51) | 51.0
  Sleep 75% 6 mo (n=55) | 20.0
  Sleep 75% 1 yr (n=53) | 28.3
  Sleep 75% 2 yr (n=51) | 17.6
  Sleep 50% 6 mo (n=55) | 18.2
  Sleep 50% 1 yr (n=53) | 5.7
  Sleep 50% 2 yr (n=51) | 17.6
  Sleep 25% 6 mo (n=55) | 7.3
  Sleep 25% 1 yr (n=53) | 15.1
  Sleep 25% 2 yr (n=51) | 7.8
  Sleep 0% 6 mo (n=55) | 10.9
  Sleep 0% 1 yr (n=53) | 11.3
  Sleep 0% 2 yr (n=51) | 5.9
  Maintain activities 100% 6 mo (n=47) | 61.7
  Maintain activities 100% 1 yr (n=44) | 65.9
  Maintain activities 100% 2 yr (n=40) | 62.5
  Maintain activities 75% 6 mo (n=47) | 19.1
  Maintain activities 75% 1 yr (n=44) | 18.2
  Maintain activities 75% 2 yr (n=40) | 17.5
  Maintain activities 50% 6 mo (n=47) | 12.8
  Maintain activities 50% 1 yr (n=44) | 0
  Maintain activities 50% 2 yr (n=40) | 15.0
  Maintain activities 25% 6 mo (n=47) | 4.3
  Maintain activities 25% 1 yr (n=44) | 9.1
  Maintain activities 25% 2 yr (n=40) | 5.0
  Maintain activities 0% 6 mo (n=47) | 2.1
  Maintain activities 0% 1 yr (n=44) | 6.8
  Maintain activities 0% 2 yr (n=40) | 0
  Transportation 100% 6 mo (n=30) | 86.7
  Transportation 100% 1 yr (n=32) | 90.6
  Transportation 100% 2 yr (n=27) | 77.8
  Transportation 75% 6 mo (n=30) | 10.0
  Transportation 75% 1 yr (n=32) | 6.3
  Transportation 75% 2 yr (n=27) | 14.8
  Transportation 50% 6 mo (n=30) | 3.3
  Transportation 50% 1 yr (n=32) | 0
  Transportation 50% 2 yr (n=27) | 0
  Transportation 25% 6 mo (n=30) | 0
  Transportation 25% 1 yr (n=32) | 0.0
  Transportation 25% 2 yr (n=27) | 3.7
  Transportation 0% 6 mo (n=30) | 0.0
  Transportation 0% 1 yr (n=32) | 3.1
  Transportation 0% 2 yr (n=27) | 3.7
  Well-being 100% 6 mo (n=22) | 54.5
  Well-being 100% 1 yr (n=24) | 58.3
  Well-being 100% 2 yr (n=17) | 47.1
  Well-being 75% 6 mo (n=22) | 31.8
  Well-being 75% 1 yr (n=24) | 33.3
  Well-being 75% 2 yr (n=17) | 35.3
  Well-being 50% 6 mo (n=22) | 9.1
  Well-being 50% 1 yr (n=24) | 0.0
  Well-being 50% 2 yr (n=17) | 11.8
  Well-being 25% 6 mo (n=22) | 4.5
  Well-being 25% 1 yr (n=24) | 8.3
  Well-being 25% 2 yr (n=17) | 5.9
  Well-being 0% 6 mo (n=22) | 0.0
  Well-being 0% 1 yr (n=24) | 0.0
  Well-being 0% 2 yr (n=17) | 0.0
  Sexual activity 100% 6 mo (n=15) | 26.7
  Sexual activity 100% 1 yr (n=14) | 57.1
  Sexual activity 100% 2 yr (n=14) | 35.7
  Sexual activity 75% 6 mo (n=15) | 33.3
  Sexual activity 75% 1 yr (n=14) | 7.1
  Sexual activity 75% 2 yr (n=14) | 14.3
  Sexual activity 50% 6 mo (n=15) | 20.0
  Sexual activity 50% 1 yr (n=14) | 14.3
  Sexual activity 50% 2 yr (n=14) | 14.3
  Sexual activity 25% 6 mo (n=15) | 20.0
  Sexual activity 25% 1 yr (n=14) | 14.3
  Sexual activity 25% 2 yr (n=14) | 28.6
  Sexual activity 0% 6 mo (n=15) | 0.0
  Sexual activity 0% 1 yr (n=14) | 7.1
  Sexual activity 0% 2 yr (n=14) | 7.1
  Employment 100% 6 mo (n=12) | 83.3
  Employment 100% 1 yr (n=12) | 75.0
  Employment 100% 2 yr (n=9) | 88.9
  Employment 75% 6 mo (n=12) | 0.0
  Employment 75% 1 yr (n=12) | 0.0
  Employment 75% 2 yr (n=9) | 0.0
  Employment 50% 6 mo (n=12) | 0.0
  Employment 50% 1 yr (n=12) | 8.3
  Employment 50% 2 yr (n=9) | 0.0
  Employment 25% 6 mo (n=12) | 0.0
  Employment 25% 1 yr (n=12) | 8.3
  Employment 25% 2 yr (n=9) | 0.0
  Employment 0% 6 mo (n=12) | 16.7
  Employment 0% 1 yr (n=12) | 8.3
  Employment 0% 2 yr (n=9) | 11.1

9. Secondary Outcome: Acetabular Insert Wear
Description: The linear wear rate of the polyethylene acetabular insert is measured radiographically and reported at 5 years.
Time Frame: 5 years
Population: Participants with available data: 97 hips were evaluated for wear rate at 5 years.
Measure: Mean (Standard Deviation); unit: millimeters per year
Units Other Than Participants: hips
Arm/Group | Accolade® TMZF® Hip Stem
Number analyzed (Participants) | 95
Number analyzed (hips) | 97
millimeters per year | 0.0342 (0.0336)
Statistical Analysis 1: Comparison: Accolade® TMZF® Hip Stem; Compare to historical control (n=94 hips): mean wear 5 years = 0.134 (0.078); Test type: Superiority or Other; p < .0001, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Wrist DXA Scan Analysis
Description: DXA is a bone densitometry scan that measures bone mineral density and assigns a T-score. This score shows the amount of bone a patient has compared with a young adult of the same gender with peak bone mass. A score above -1 is considered normal. A score between -1 and -2.5 is classified as osteopenia (low bone mass). A score below -2.5 is defined as osteoporosis.
Time Frame: 5 years
Population: Participants with available data: 107 hips had DXA scan T-scores at 5 years.
Measure: Mean (Standard Deviation); unit: T-score
Units Other Than Participants: hips
Arm/Group | Accolade® TMZF® Hip Stem
Number analyzed (Participants) | 105
Number analyzed (hips) | 107
T-score | -0.4 (1.05)
Statistical Analysis 1: Comparison: Accolade® TMZF® Hip Stem; Compare Wrist DXA T-score preop to 5 years; Test type: Superiority or Other; p = .0002, Sign test

ADVERSE EVENTS:
Time Frame: This study requires that all operative site and serious systemic adverse events be reported from enrollment to 5 years postoperative. Censored protocol violations were not included as at risk participants.
Description: Elective procedures not included.e.g.non-study joint replacement/revision,rotator cuff repair,carpal tunnel release,cataract,intra-ocular & bunion procedures,total shoulder repair,laminectomy,microdiscectomy,breast reduction,cervical spine fusion,& mid/flat-foot surgery. Industry standard AE terms not used; specific AE terms not used for all AEs
Groups:
- Accolade TMZF Hip Stem: Participants who received the Accolade TMZF Hip Stem
Arm/Group | Accolade TMZF Hip Stem
Serious Adverse Events (participants affected / at risk) | 65/234
Other Adverse Events (participants affected / at risk) | 54/234
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Accolade TMZF Hip Stem (N=234)
Non-operative site (Blood and lymphatic system disorders) | 2 (2)
Non-operative site (Cardiac disorders) | 10 (13)
Non-operative site (Endocrine disorders) | 1 (1)
Non-operative site (Gastrointestinal disorders) | 7 (7)
Non-operative site (General disorders) | 4 (4)
Non-operative site (Infections and infestations) | 2 (2)
Operative site (Infections and infestations) | 2 (2)
Non-operative site (Injury, poisoning and procedural complications) | 2 (2)
Operative site (Injury, poisoning and procedural complications) | 3 (3)
Non-operative site (Musculoskeletal and connective tissue disorders) | 8 (8)
Operative site (Musculoskeletal and connective tissue disorders) | 16 (18)
Non-operative Site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (7)
Non-operative site (Nervous system disorders) | 3 (3)
Non-operative site (Renal and urinary disorders) | 3 (3)
Non-operative site (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Non-operative site (Skin and subcutaneous tissue disorders) | 1 (1)
Non-operative site (Vascular disorders) | 6 (8)
Operative site (Nervous system disorders) | 1 (1)
Non-operative site (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Accolade TMZF Hip Stem (N=234)
Operative site Musculoskeletal and Connective tissue disorders (Musculoskeletal and connective tissue disorders) | 54 (63)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Each investigator shall have privileges for their own center's results at the completion of the study. These manuscripts and abstracts will be delayed until after the multi-center publication is submitted.All publications shall be submitted to the sponsor for review at least 60 days prior to submission for publication.The sponsor shall not edit or otherwise influence the publications other than to ensure that confidential information is not disclosed and that the data is accurately represented.